CLINICAL TRIAL: NCT00902655
Title: Desmopressin in the Treatment of Mixed Nocturia With Nocturnal Polyuria and Low Nocturnal Bladder Capacity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-04-05
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Nocturia
Keywords: Nocturnal polyuria; Nocturnal bladder capacity
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin (Experimental)
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Desmopressin 0.1,0.2 or 0.4 mg once daily for 3-weeks of dose titration phase and 4-weeks of treatment phase
  Other Names: Minirin

SUMMARY:
Nocturia is defined as waking one or more times to void during the period between going to bed with the intention of sleeping and waking with the intention of arising.The pathophysiology of nocturia is multifactorial and can be complex. Therefore it is important to adopt a systematic approach to identify the possible causal factors of nocturia and to treat them accordingly. Patients with nocturia can be categorized as having one of the following three disorders: (1) nocturnal polyuria (NP) in which the voided urine volume during the hours of sleep exceeds 35% of the 24-hr output, (2) low nocturnal bladder capacity (NBC) causing a nocturnal urinary volume greater than the bladder capacity, (3) or mixed nocturia, a combination of the preceding two categories.

Desmopressin, a synthetic analogue of the antidiuretic hormone (ADH), has been used for many years to treat diabetes insipidus and primary nocturnal enuresis.More recently, it is also known to be effective against nocturia with NP by decreasing night-time urine production.However, it may be associated with an increased risk of developing hyponatremia due to water retention, especially in elderly patients.In the present study, we investigated the safety and efficacy of oral desmopressin for the treatment of mixed nocturia in patients with both NP and a low NBC.

DETAILED DESCRIPTION:
1. Open label, prospective, multicenter study
2. Study design

   * screening (1-week), dose titration (1-3 weeks) and 4-weeks of treatment period
   * open-label dose-titration periods of up to 3 wk; the patients' optimum oral desmopressin dose (0.1, 0.2 and 0.4 mg) was determined as the dose that decreased the number of nocturnal voids by ≥50% and NUV decreased by ≥20% without hyponatremia.
   * If the patients did not meet the above criteria during dose titration period, they received the maximum tolerable dose instead of the optimum dose. -- 4-weeks of treatment period; Eligible patients were treated with the determined optimum desmopressin dose for 4-weeks.
3. Measurements

   * 3-day frequency-volume charts
   * sleep questionnaire
   * body weight, blood and urine analysis,serum sodium monitoring
   * adverse event

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 yr
* nocturia ≥2 voids/night
* nocturnal polyuria index (NPi) >33%
* nocturnal bladder capacity index (NBCi) >1

Exclusion Criteria:

* nocturia due to other defined causes of increased urinary frequency
* primary polydipsia (>40mL/kg/24 h)
* neurogenic bladder dysfunction
* significant bladder outlet obstruction
* urge incontinence
* continued post-voiding residual urine >150mL
* serum sodium levels <135mmol/L
* uncontrolled hypertension characterized by fluid and/or electrolyte imbalance
* use of diuretics
* actual or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a 50% or greater reduction in the mean number of nocturnal voids compared with baseline levels. | after 4-weeks of treatment phase

SECONDARY OUTCOMES:
Change in the mean number of nocturnal voids. | after 4-weeks of treatment phase
Change in the mean duration of the period from bedtime to the first nocturnal void. | after 4-weeks of treatment phase
Change in the proportion of patients that felt they had a good sleep experience. | after 4-weeks of treatment phase
Body weight gain. | after 4-weeks of treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (6):
- South Korea (6):
  - Keimyung University School of Medicine, Daegu
  - College of Medicine Inha University, Inchon
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University College of Medicine, Seoul